CLINICAL TRIAL: NCT07044570
Title: Using Real-Time Data Capture to Examine Implicit Attitudes as Mediators of Physical Activity Adherence in Interventions
Brief Title: eMOTION: Examining Implicit Attitudes in Physical Activity Engagement
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Genevieve Dunton, Chief, Division of Health Behavior Research and Director, USC Real-Time Eating Activity and Children's Health (REACH) Lab, University of Southern California
Other Study IDs: UP-24-00381; R03CA292977 (NIH)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Physical Activity; Overweight or Obesity; Cancer
Keywords: Affective Response; Psychological Needs; Physical Activity; Implicit Attitudes
MeSH Terms: conditions — Motor Activity; Overweight; Obesity; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Affect (no enhancements) > Intensity: Participants receive affect-based goals for the first 8-weeks, then cross-over to receive intensity-based goals for the second 8-weeks. No enhancements are added to the standard mHealth intervention.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention
- Intensity > Affect (no enhancements): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. No enhancements are added to the standard mHealth intervention.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention
- Affect (+ SAVOR + TYPE/CONTEXT) > Intensity: Participants receive affect-based goals for the first 8-weeks. In addition to the standard mHealth intervention, participants engage in both SAVOR and TYPE/CONTEXT enhancements to augment the treatment effects of the affect-based goals condition. Participants then cross-over to receive intensity-based goals for the second 8-weeks.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement; Behavioral: SAVOR enhancement
- Intensity > Affect (+ SAVOR + TYPE/CONTEXT): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. In addition to the standard mHealth intervention, participants engage in both SAVOR and TYPE/CONTEXT enhancements to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement; Behavioral: SAVOR enhancement
- Affect (+SAVOR) > Intensity: Participants receive affect-based goals for the first 8-weeks. In addition to the standard mHealth intervention, participants engage in the SAVOR enhancement to augment the treatment effects of the affect-based goals condition. Participants then cross-over to receive intensity-based goals for the second 8-weeks.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: SAVOR enhancement
- Intensity > Affect (+SAVOR): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. In addition to the standard mHealth intervention, participants engage in the SAVOR enhancement to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: SAVOR enhancement
- Affect (+TYPE/CONTEXT) > Intensity: Participants receive affect-based goals for the first 8-weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT enhancement to augment the treatment effects of the affect-based goals condition. Participants then cross-over to receive intensity-based goals for the second 8-weeks.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement
- Intensity > Affect (+TYPE/CONTEXT): Participants receive intensity-based goals for the first 8-weeks, then cross-over to receive affect-based goals for the second 8-weeks. In addition to the standard mHealth intervention, participants engage in the TYPE/CONTEXT enhancement to augment the treatment effects of the affect-based goals condition.
  Interventions: Behavioral: Physical Activity Goals mHealth Intervention; Behavioral: TYPE/CONTEXT enhancement

INTERVENTIONS:
Behavioral: Physical Activity Goals mHealth Intervention — On days participants plan to exercise, they engage in two daily goal sessions (morning and evening). Morning sessions provide an activity goal for the day and ask the participant to create a plan, anticipate barriers, and brainstorm solutions for achieving this goal. The affect-based goal condition asks participants to engage in either (1) a type (50% of daily goals) or (2) a context (50% of daily goals) of physical activity that allows them to experience positive affect. Goals focused on context are randomly generated to suggest that the participant performs activity (1) in a place; (2) in a social situation; or (3) while listening to something that makes them feel good. The intensity-based goal condition asks participants to maintain a certain target heart rate range during physical activity. Starting heart rate reflects the approximate age-adjusted heart rate max, with goals progressively increasing from 55% to 70% heart rate max.
Behavioral: TYPE/CONTEXT enhancement — TYPE/CONTEXT augments intervention effects by providing tailored recommendations for activity types and contexts that satisfy personally-important psychological needs as rated by each participant at baseline. Ratings from a crowdsourced panel of adults on Amazon Mechanical Turk will be used to determine the potential for specific activity types and contexts to satisfy psychological needs; our tailoring algorithm will then recommend the corresponding activity type or context while accounting for reported constraints (e.g., ability, access). These details will be incorporated into a tailored recommendation provided to participants each Sunday as they make activity plans for the upcoming week. Specifically, the program will randomly select either type or context (i.e., location, audio, social) recommendations and will rotate every two weeks. For TYPE, participants' top 3 activity types are recommended; for CONTEXT, participants' top 3 activity contexts are recommended.
  Groups: Affect (+ SAVOR + TYPE/CONTEXT) > Intensity; Affect (+TYPE/CONTEXT) > Intensity; Intensity > Affect (+ SAVOR + TYPE/CONTEXT); Intensity > Affect (+TYPE/CONTEXT)
Behavioral: SAVOR enhancement — SAVOR implements a brief savoring exercise on the smartphone that takes place either after the planned physical activity session or during the evening goal session (after the self-monitoring module). Participants will respond to questions that are intended to enhance and prolong positive experiences during physical activity. To trigger attentional deployment, a common savoring strategy that involves intensifying experiences by focusing on them, participants will answer three open-ended prompts. These prompts are drawn from a prompt pool with slightly varied wording to promote a sense of novelty. Savoring prompts will rotate daily and have a day lag built in every week (i.e., Week 1 Monday Savoring Prompts are Week 2 Tuesday Savoring Prompts).
  Groups: Affect (+ SAVOR + TYPE/CONTEXT) > Intensity; Affect (+SAVOR) > Intensity; Intensity > Affect (+ SAVOR + TYPE/CONTEXT); Intensity > Affect (+SAVOR)

SUMMARY:
This early-phase trial will test intervention strategies to influence implicit attitudes towards physical activity and determine whether changes in those mechanisms result in change in physical activity behavior among inactive adults who are overweight or obese.

DETAILED DESCRIPTION:
This ORBIT model phase 1 trial will examine whether implicit attitudes (1) can be experimentally manipulated in real-world settings; and (2) mediate the relationship between interventions and physical activity behavior. A novel physical activity intervention will be optimized by efficiently disentangling the effects of its core component and two enhancement components on affective mechanisms associated with physical activity engagement.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Reside in the United States
3. Self-reported BMI ≥ 25
4. Current structured physical activity engagement < 60 minutes per week
5. Own a personal smartphone device
6. Reside in an area with Internet or Wi-Fi connectivity during the study period
7. Able to speak and read in English
8. Interested and willing to start a physical activity program
9. Willing to wear a Fitbit Versa smartwatch provided by the study team everyday continuously (including at work and during physical activity), in place of any Fitbits or smartwatches previously worn, for the duration of the study period
10. Able to read the small font on a smartwatch screen without glasses, or willing to carry reading glasses during physical activity for the purpose of reading the smartwatch screen
11. Enrolled in the parent eMOTION intervention study

Exclusion Criteria:

1. Inability to provide informed consent due to cognitive disability
2. Inability to engage in one or more key treatment components, including those with medical conditions that preclude physical activity engagement or who cannot wear an accelerometer on the wrist or answer brief surveys on the smartwatch for any reason
3. Current pregnancy
4. Referred to the study by another participant or from Reddit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physically inactive adults with overweight or obesity who are living in the U.S.,
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Implicit Attitudes | Up to once daily for weeks 2-9 and weeks 12-19
  The single-category Implicit Association Test (IAT) will ask participants to match to a conceptual target such as sedentary behavior (e.g., sitting, lying) or physical activity (e.g., walking, running) to affective attributes (e.g., good/bad).If the participant has a strong automatic association between the attribute and conceptual target, then the reaction time will be shorter (representing a favorable implicit attitude). A real-time audibly prompted IAT will be triggered on participants' smartphones in the morning on days a physical activity session is planned (with four reminders sent once every hour if incomplete).

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve F Dunton, PhD MPH, Principal Investigator — University of Southern California
Locations (1):
- Univeristy of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No